CLINICAL TRIAL: NCT04521114
Title: A Phase II, Multi-center, Two-Part, Three-Arm, Dose-Ranging Study of the Safety and Efficacy of Leronlimab (PRO 140) in Adult Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Leronlimab (PRO 140) in Patients With Nonalcoholic Steatohepatitis
Acronym: NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDI-NASH-01
Record Dates: First submitted 2019-11-18; First posted 2020-08-20 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: NASH; PRO 140; Leronlimab
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Leronlimab 700 mg (Experimental): Leronlimab 700 mg SC weekly injection
  Interventions: Drug: leronlimab 700 mg
- Leronlimab 350 mg (Experimental): Leronlimab 350 mg SC weekly injection
  Interventions: Drug: leronlimab 350 mg
- Placebo (Placebo Comparator): Placebo SC weekly injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo will be administered subcutaneously every week for 13 weeks.
  Arms: Placebo
Drug: leronlimab 700 mg — 700 mg leronlimab will be administered subcutaneously every week for 13 weeks.
  Other Names: PRO 140
  Arms: Leronlimab 700 mg
Drug: leronlimab 350 mg — 350 mg leronlimab will be administered subcutaneously every week for 13 weeks.
  Other Names: PRO 140
  Arms: Leronlimab 350 mg

SUMMARY:
This is a phase II study of of Leronlimab (PRO 140)-Humanized monoclonal antibody to CCR5 in patients with Nonalcoholic Steatohepatitis (NASH).

DETAILED DESCRIPTION:
This is an exploratory phase II, multi-center, two-part study (Part 1: randomized, placebo-controlled, two-arm with 60 patients; Part 2: non-randomized, single-arm, open-label with 30 patients) designed to evaluate the safety and efficacy of leronlimab after subcutaneous (SC) administration in patients with NASH for 13 weeks.

A Follow Up visit was conducted 28 (± 3) days after receiving the last study treatment (i.e., after last dose of Leronlimab (PRO 140) or placebo.

ELIGIBILITY:
Inclusion Criteria: Subjects are required to meet ALL of the following criteria for enrollment into the study:

1. Subject is a male or female between 18 to 75 years of age inclusive.
2. Evidence of nonalcoholic steatohepatitis (NASH) based on one of the following criteria:

   * Criteria 1: Histologically-confirmed diagnosis of NASH on a liver biopsy, or
   * Criteria 2: FibroScan or Shearwave US during screening (or within 6 months before screening) shows kPa ≥7 but <14 and CAP ≥260.
3. Subject shows presence of hepatic fat fraction as defined by ≥ 8% on MRI-PDFF and cT1 ≥ 800 ms at Screening.
4. Has had a stable body weight (±5%) within 6 months prior to Screening.
5. Body Mass Index (BMI) ≥ 28 kg/m2 at Screening
6. Has clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
7. Laboratory Screening results as indicated below:

   1. AST:ALT Ratio ≤ 1, if AST or ALT value is > ULN
   2. Screening Liver enzymes (AST, ALT, and ALK PHOS) < 5 x ULN.
   3. Total Bilirubin ≤ 1.3 mg/dL (except if Gilbert's Disease)
   4. Platelet count ≥ 150,000/mm3
   5. International normalized ratio (INR) < 1.3
   6. Estimated Glomerular Filtration Rate (eGFR) ≥ 60/mL/min
   7. Glycosylated hemoglobin (HbA1c) < 9%.
   8. Thyroid-Stimulating Hormone (TSH) within normal reference range. Note: Any subject with a non-clinically significant TSH value outside of the normal range may be enrolled if their T3 and free T4 values are within the normal range.
8. Subjects with pre-diabetes or type 2 diabetes will be allowed to participate if the following criteria is met:

   * Subjects who are taking anti-diabetic medications should be on a stable dose for a period of at least 3 months prior to Screening and do not anticipate clinically significant dose adjustments during the course of study.
   * Subjects must be on a stable diet/lifestyle regimen for at least 3 months prior to screening and do not anticipate a clinically significant change during the course of study.
9. Subjects who are taking Vitamin E should be on a stable dose of Vitamin E (if ≥ 400 IU) for a period of at least 4 weeks prior to Screening and do not anticipate dose adjustments for the duration of the study.
10. Both male and female patients and their partners of childbearing potential must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, tubal sterilization or vasectomy) or must practice complete abstinence from intercourse of reproductive potential from study entry to 6 months after the last day of treatment (excluding women who are not of childbearing potential and men who have been sterilized).
11. Females of child-bearing potential must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and Male participants must agree to use contraception and refrain from donating sperm for at least 90 days after the last dose of study intervention.
12. Subject is willing and able to give informed consent prior to any study specific procedures being performed.
13. Subject is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures and study restrictions

Exclusion Criteria: Subjects meeting ANY of the following criteria will be excluded from enrollment:

1. Any concurrent clinically significant liver disease with an etiology other than NASH including autoimmune hepatitis, alcoholic hepatitis, hypoxic/ischemic hepatopathy, and biliary tract disease.
2. History of alcohol consumption greater than 21/units/week (for males) and 14/units/week (for females) within the last 2 years prior to screening.

   Note: Use of online unit calculator for alcohol consumption is recommended (e.g., https://alcoholchange.org.uk/alcohol-facts/interactive-tools/unit-calculator)
3. Any drug-induced steatohepatitis secondary to amiodarone, corticosteroids, estrogens, methotrexate, tetracycline, or other medications known to cause hepatic steatosis.
4. Undergone major surgery, including liver surgery, within 6 months prior to screening deemed clinically significant by the investigator.
5. Prior or pending liver transplantation.
6. History or presence of cirrhosis or stage 4 fibrosis in historical liver biopsy and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding.
7. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test), hepatitis C (defined as having a positive Anti-HCV test with detectable reflex HCV RNA; Note: Subject with positive Anti-HCV test and with undetectable HCV RNA would not be excluded), acute hepatitis A (defined as subjects with serum positive for hepatitis A IgM (HAV) antibody) or acute hepatitis E (defined as having anti-HEV IgM antibody).
8. Any active infection requiring systemic therapy at the time of screening, which is considered clinically significant per the Investigator.
9. Positive test for human immunodeficiency virus (HIV) or HIV infection.
10. History of bleeding diathesis within 6 months of screening.
11. Any malignancy within the past 5 years, excluding successfully treated basal cell carcinoma or squamous cell carcinoma without evidence of metastases.
12. Seizure disorder requiring ongoing antiseizure therapy or with any condition that, in the judgment of the investigator, is likely to increase the risk of seizure (e.g. CNS malignancy)
13. Clinically significant active cardiac disease which would interfere with study conduct or study results interpretation per the PI.
14. Any known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Prior therapy with Leronlimab or any other CCR5 antagonist (e.g. maraviroc) within 6 months prior to screening.
16. History of severe allergic, anaphylactic, or other hypersensitivity reactions to humanized monoclonal antibodies.
17. Any condition requiring continuous systemic treatment with immunosuppressive (such as corticosteroids) or immunomodulatory medications.

    Note: Inhaled or topical steroids of up to 5 mg daily prednisone equivalent dose are permitted in the bsence of active autoimmune disease.
18. History of administration of a live, attenuated vaccine within four weeks prior to start of PRO 140 treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study.

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed. However intranasal influenza vaccines (e.g., Flu-Mist ®) are live attenuated vaccines, and are not allowed.
19. Currently participating in an investigational study or received an investigational drug within 28 days or 5 half-lives (whichever is longer) prior to study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Southern California Research Center, Coronado, California
  - Meridien Research, Maitland, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Care United Research LLC, Forney, Texas
  - American Research Corporation, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munteanu M, Tiniakos D, Anstee Q, Charlotte F, Marchesini G, Bugianesi E, Trauner M, Romero Gomez M, Oliveira C, Day C, Dufour JF, Bellentani S, Ngo Y, Traussnig S, Perazzo H, Deckmyn O, Bedossa P, Ratziu V, Poynard T; FLIP Consortium and the FibroFrance Group. Diagnostic performance of FibroTest, SteatoTest and ActiTest in patients with NAFLD using the SAF score as histological reference. Aliment Pharmacol Ther. 2016 Oct;44(8):877-89. doi: 10.1111/apt.13770. Epub 2016 Aug 23. PMID 27549244
- See also: Diagnostic performance of FibroTest — https://pubmed.ncbi.nlm.nih.gov/27549244/

RESULTS

PARTICIPANT FLOW:
Groups:
- Leronlimab 700 mg: 700 mg SC weekly injection
- Leronlimab 350 mg: 350 mg SC weekly injection
Period: Overall Study
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Started | 30 | 27 | 30
Completed | 24 | 21 | 28
Not Completed | 6 | 6 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Sponsor Wish | 1 | 0 | 0
Not completed — Withdrawal of Consent | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Patients with Nonalcoholic Steatohepatitis (NASH)
Groups:
- Leronlimab 700 mg: 700mg SC weekly injection
- Leronlimab 350 mg: 350mg SC weekly injection
- Total: Total of all reporting groups
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo | Total
Number analyzed (Participants) | 30 | 27 | 30 | 87
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 53.2 (13.68) | 52.4 (8.38) | 55.6 (10.47) | 53.80 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 9 | 41
  Male | 11 | 14 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 12 | 44
  Not Hispanic or Latino | 14 | 11 | 18 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 2 | 7
  White | 30 | 22 | 28 | 80
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 41.2 (9.56) | 38.0 (5.52) | 38.4 (5.89) | 39.2 (7.33)

OUTCOME MEASURES:

1. Primary Outcome: MRI-PDFF Change From Baseline to Week 14
Description: Change in hepatic fat fraction from baseline assessed by magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) at week 14
Time Frame: Change from baseline (day one, first day of treatment) to EOT (day 92, 13 weeks of treatment)
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Percentage of hepatic fat fraction
Groups:
- Leronlimab 350 mg: Leronlimab 350mg SC weekly injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 28
Percentage of hepatic fat fraction | -1.25 [-2.60 to 2.30] | -0.90 [-3.10 to 0.40] | 0.90 [-0.20 to 3.70]

2. Secondary Outcome: MRI-cT1 Change From Baseline to Week 14
Description: MRI corrected T1 (cT1) is emerging as a promising quantitative surrogate metric for assessing a composite of liver inflammation and fibrosis.
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Milliseconds (ms)
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 28
Milliseconds (ms) | -7.0 [-35.0 to 22.0] | -2.00 [-54.00 to 24.00] | 22.0 [2.0 to 41.0]

3. Secondary Outcome: Alkaline Phosphatase
Description: Change from Baseline to Week 14 in Alkaline Phosphatase
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Leronlimab 700 mg: Leronlimab 700 mg SC weekly injection
  .
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
IU/L | 0.37 (7.77) | -3.68 (7.99) | -0.83 (7.75)

4. Secondary Outcome: Alanine Aminotraferase (ALT)
Description: Change from Baseline to Week 14 in Alanine Aminotraferase (ALT)
Time Frame: Measured at baseline (day 1) and at day 92
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
U/L | 4.77 (32.06) | -0.76 (16.65) | 1.79 (18.83)

5. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: Change from Baseline to Week 14 in Aspartate Aminotransferase (AST)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Leronlimab 700 mg: Leronlimab (700mg) SC weekly injection
  .
- Leronlimab 350 mg: Leronlimab (350 mg) SC weekly injection
- Placebo: Placebo (0 mg) SC weekly injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
U/L | 1.40 (15.10) | -6.12 (33.33) | 2.17 (13.23)

6. Secondary Outcome: GGT S
Description: Change from Baseline to Week 14 in Gamma Glutamyl transferase, GGT S
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Leronlimab 700 mg: Leronlimab (700mg) SC weekly injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
U/L | 5.67 (14.12) | -3.00 (14.73) | 0.90 (11.61)

7. Secondary Outcome: Neutrophils/Leukocytes
Description: Change in Neutrophils/Leukocytes ratio from Baseline to Week 14
Time Frame: Measured at baseline (day 1, start of treatment) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio of neutrophils to leukocytes
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
Ratio of neutrophils to leukocytes | 0.93 (5.94) | -4.32 (8.42) | 0.55 (6.07)

8. Secondary Outcome: CCL2
Description: Change from Baseline to Week 14 in Monocyte Chemotactic Protein 1 (CCL2)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 57.60 (175.98) | -77.0 (161.99) | -38.57 (140.75)

9. Secondary Outcome: CCL3
Description: Change from Baseline (day 1, start of treatment) to Week 14 (EOT) in Macrophage Inflammatory Protein 1 Alpha
Time Frame: Measured at baseline (day 1, start of treatment) and at EOT (day 92)
Population: Safety Analysis Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 1.40 (6.22) | -7.20 (5.03) | -0.96 (2.62)

10. Secondary Outcome: CCL5 (Rantes)
Description: Change from Baseline to Week 14 in CCL-5 (Rantes)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: Placebo SC injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
ng/mL | 8.14 (15.82) | -6.80 (44.40) | -0.39 (8.28)

11. Secondary Outcome: Fibro Test Score
Description: Change from baseline (day 1, start of treatment) to Week 14 (EOT) in Fibro Test Score measured on a scale of 0 to 1, where 0 to 0.27 is no fibrosis, 0.27 to 0.48 is minimal fibrosis, 0.48 to 0.58 is moderate fibrosis, 0.58 to 0.74 is advanced fibrosis and 0.74 to 1.00 is severe fibrosis (Cirrhosis). Minimum score is zero, maximum score (worst outcome) is 1.
Time Frame: Measured at baseline (day 1, start of treatment) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Leronlimab 700 mg: Leronlimab 700 mg SC injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29
score on a scale | 0.02 (0.06) | 0.01 (0.07) | -0.00 (0.06)

12. Secondary Outcome: CCL11( Eotaxin-1)
Description: Change from Baseline to Week 14 in Eosinophils Chemotactic Protein
Time Frame: Measured at baseline (day 1, start of treatment) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 29.30 (87.67) | -3.88 (95.10) | -41.32 (116.25)

13. Secondary Outcome: CCL18
Description: Change from Baseline to week 14 in CCL18 (Pulmonary & Activation-Reg Chemokine)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
ng/mL | 6.77 (36.16) | -27.28 (40.49) | -2.14 (34.43)

14. Secondary Outcome: VCAM
Description: Change from Baseline to Week 14 in Vascular Cell Adhesion Molecule 1
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Leronlimab 700 mg: Leronlimab 700 mg weekly injection
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
ng/mL | 35.93 (178.64) | -82.80 (79.95) | 8.89 (109.96)

15. Secondary Outcome: Interleukin-1 Beta
Description: Change from Baseline to Week 14 in Interleukin-1 Beta
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 0.06 (0.31) | 0.09 (0.46) | 0.16 (0.61)

16. Secondary Outcome: IL-1RA
Description: Change from Baseline to Week 14 in Interleukin 1 Receptor Antagonist
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Leronlimab 700 mg: Leronlimab 700mg SC weekly injection
- Placebo: Placebo (Randomized)
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 6.37 (125.39) | -16.24 (74.40) | 15.93 (54.63)

17. Secondary Outcome: IL-6
Description: Change from Baseline to Week 14 in Interleukin 6
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 0.17 (1.18) | -0.24 (0.68) | 0.31 (1.74)

18. Secondary Outcome: IL-8
Description: Change from Baseline to Week 14 in Interleukin 8
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | -3.25 (8.89) | -2.18 (7.81) | -0.54 (5.00)

19. Secondary Outcome: TNF Receptor 2
Description: Change from baseline (day 1, start of treatment) to Week 14 (EOT) in Tumor Necrosis Factor Receptor 2
Time Frame: Measured at baseline (day 1, start of treatment) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
pg/mL | 1.04 (3.25) | -1.66 (2.24) | 0.79 (1.72)

20. Secondary Outcome: TIMP-1
Description: Change from Baseline (day 1, start of treatment) to Week 14 (EOT) in Tissue Inhibitor of Metalloproteinases 1 (ng/mL)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Leronlimab 350 mg: Leronlimab 350 mg (Non-Randomized)
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
ng/mL | 8.30 (32.39) | -11.76 (29.33) | 1.25 (25.62)

21. Secondary Outcome: En Rage
Description: Change from baseline (start of treatment, day 1) to Week 14 (EOT) in En Rage (Receptor Advanced Glycation End-Products)
Time Frame: Measured at baseline (day 1) and at EOT (day 92)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 28
ng/mL | 30.77 (229.87) | -60.40 (245.32) | 54.96 (141.75)

ADVERSE EVENTS:
Time Frame: 14 Weeks
Groups:
- Leronlimab 700 mg: Leronlimab 700mg (Randomized)
Arm/Group | Leronlimab 700 mg | Leronlimab 350 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 1/27 | 2/30
Other Adverse Events (participants affected / at risk) | 28/30 | 21/27 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab 700 mg (N=30) | Leronlimab 350 mg (N=27) | Placebo (N=30)
TOOTH ABSCESS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
EYE INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — One death was based on a car accident and was not believed to be related to treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leronlimab 700 mg (N=30) | Leronlimab 350 mg (N=27) | Placebo (N=30)
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2
C-reactive protein increased (Investigations) | 7 | 8 | 3
Abdominal Pain (Gastrointestinal disorders) | 5 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 2
Urinary tract infection (Renal and urinary disorders) | 5 | 3 | 3
Injection site erythema (General disorders) | 2 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2 | 2
Injection site pain (Injury, poisoning and procedural complications) | 3 | 1 | 2
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hyperglycaemia (Endocrine disorders) | 4 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 1
Hypertension (Vascular disorders) | 2 | 3 | 1
Injection site pruritus (Gastrointestinal disorders) | 2 | 1 | 2
COVID-19 (Infections and infestations) | 2 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04521114/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04521114/SAP_001.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04521114/ICF_002.pdf